CLINICAL TRIAL: NCT01403649
Title: Strategies to Vaccinate All Children for Influenza in a Practice Setting
Brief Title: Collaborative Efforts to Increase Flu Vaccination
Acronym: CollabFlu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-0589; 1U01IP000320 (NIH)
Record Dates: First submitted 2011-07-14; First posted 2011-07-27 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Influenza; Collaboration
MeSH Terms: conditions — Influenza, Human | interventions — Patients' Rooms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increasing flu vaccination (Experimental): Collect from billing records in the 10 intervention practice sites to test for an increase in the rate of receipt of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children 6 months to 18 years during the season. The interventions include: 1. Develop practice-based intervention strategies (like use of reminder-recall of children due for influenza,2. Develop Private/public collaboration to increase flu vaccination between the intervention practices, their county public health department and visiting nursing associations, and 3. Implement both practice-based and private-public collaborative strategies in the intervention practices while monitoring only in the control practices
  Interventions: Behavioral: Private/public collaboration to increase flu vaccination
- Usual care (Other): Patients in control practices will continue to receive usual care with no change in practice regarding influenza immunization delivery.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Private/public collaboration to increase flu vaccination — Intervention practices will develop office-based interventions including methods to identify high-risk patients within their practices and methods of maximizing the immunization of these children within the practice, use of patient reminders, after-hours influenza clinics, walk-in provision of influenza vaccine and increased focus on education regarding the need for immunization. The practices will also collaborate with their county public health departments and visiting nursing associations to develop private-public collaborative interventions that may include large clinics for school-aged children for multiple practices and tracking of influenza supplies and redistribution of influenza vaccine between practices when supplies are delayed or inadequate.
  Arms: Increasing flu vaccination
Other: Usual care — This group will continue administering influenza vaccine to their patients in their practice as they normally do.
  Arms: Usual care

SUMMARY:
Beginning with the 2009-2010 season, influenza vaccine is universally recommended for children age 6 months to 18 years old, placing extra burden on health care providers across the U.S. The focus of this study is to develop new strategies and implement existing evidence-based strategies to enhance influenza immunization in these children. The intervention will involve collaboration from different types of primary care providers, the Colorado Immunization Information System (CIIS), public health departments and visiting nursing services (VNA). It will be designed and implemented by those involved with delivery with a focus on sustainability after the completion of the study. Parental input will be gathered during the planning year through focus groups to assist in developing the intervention. Qualitative assessments and examination of processes during the first year of implementation will guide modifications during the second implementation year in order to assure sustainability. Primary outcome measures in the intervention and control groups: 1) increase in the rate of receipt of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children 6 mo.-18 yr. and 2) increase in the rate of children 6 mo.-18 yr. who were fully immunized (received all required influenza injections) during the season. 3) measure outcomes by age group (6 mo.-5 yr., 6-8 yr., 9-12 yr., 13-18 yr.) and types of clinical sites (urban Peds, urban FM, rural FM)

DETAILED DESCRIPTION:
Specific Aim 1: Within each of three types of clinical sites (urban pediatric, urban family medicine, and rural family medicine) recruit a group of similar practices (Year 1) 1a. Randomize practices within each type of clinical site to either the intervention or the control group

1b. Establish private-public collaborations for influenza vaccination delivery between county public health departments, visiting nursing associations and each of the intervention practices within the three clinical site types

Specific Aim 2: Conduct focus groups among parents of children seen at intervention practices, to assess attitudes and perceived barriers to possible practice-based and collaborative strategies to promote influenza vaccination (Year 1)

Specific Aim 3: Develop (Year 1) and implement (Years 2 and 3) a plan for comprehensive and collaborative delivery of influenza vaccine at intervention practices 3a. Develop practice-based intervention strategies focusing primarily on immunization of high-risk patients 3b. Develop private-public collaborative interventions between the intervention practices, their county public health department and visiting nursing associations focusing primarily on immunization of school-aged children 3c. Implement (Years 2 and 3) both practice-based and private-public collaborative strategies in the intervention practices while monitoring only in the control practices

Specific Aim 4: Conduct a group-randomized trial to evaluate and compare the effectiveness of the comprehensive delivery model in improving influenza vaccination coverage for children 6 months to 18 years in three different types of clinical sites (urban pediatric, urban family medicine, and rural family medicine).

4a. Evaluate effectiveness of the comprehensive delivery model at each of the three types of clinical sites

1. Compare the following primary outcome measures in the intervention and control groups: 1) increase in the rate of receipt of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children 6 months to 18 years and 2) increase in the rate of children 6 months to 18 years who were fully immunized (received all required influenza injections) during the season.
2. Compare the following secondary outcome measures: 1) increase in the rate of receipt of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among high-risk children and 2) increase in the rate of high-risk children who were fully immunized during the season.
3. Evaluate sustainability of the comprehensive delivery model on the above outcome measures

4b. Compare the effectiveness of the comprehensive delivery model in three different types of clinical sites (urban pediatric private practice, urban family medicine private practice, and rural family medicine private practice)

Specific Aim 5: Evaluate the process of implementation of the comprehensive delivery model for influenza delivery in each of the three types of sites.

5a. Assess process measures relevant to implementation of practice-based interventions and compare by type of clinical site 5b. Assess process measures relevant to implementation of private-public collaborative interventions and compare by type of clinical site 5c. Using key informant interviews, assess perceptions regarding facilitators and barriers to private-public collaborative delivery, alternative methods and means of improving the process among practice providers, administrators and among participating public health and visiting nurse personnel

Specific Aim 6: In two urban pediatric intervention practices and one rural family medicine practice, conduct surveys examining parental attitudes about methods of influenza delivery and their experience with their practice's participation in a comprehensive and collaborative private-public model for influenza delivery

Major Hypotheses:

SA4. Hypothesis 1. Effectiveness on receipt of ≥1 influenza vaccine: The increase in the likelihood of receiving ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children 6 months to 18 years will be greater for children in intervention practices than in control practices.

SA4. Hypothesis 2 Effectiveness - fully immunized: The increase in the likelihood of receiving all necessary influenza vaccines during the post-intervention year compared to the pre-intervention year among children 6 months to 18 years will be greater for children in intervention practices than in control practices.

SA4. Hypothesis 3. Effectiveness by age strata: The increase in the likelihood of receiving ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children in each of the following age strata will be greater in intervention than in control practices: 1) 6 months through 5 years; 2) 6 through 8 years; 3) 9 through 12 years; 4) 13 through 18 years.

SA4. Hypothesis 4. Effectiveness in high-risk children: The increase in the likelihood of receiving of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among high-risk children 6 months to 18 years will be greater for high-risk children in intervention practices than in control practices.

SA4. Hypothesis 5. Sustainability: The increase in the likelihood of receiving ≥1 influenza vaccine during the second post-intervention year compared to the pre-intervention year among children 6 months to 18 years will be greater for children in intervention practices than in control practices. (Sustainability will also be evaluated for other outcomes above.)

SA4. Hypothesis 6. Differential effectiveness by clinical site type: The increase in the likelihood of receiving of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among children 6 months to 18 years for intervention vs. controls will differ by clinical site type

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 mo - 18 yr in up to 20 practices

Exclusion Criteria:

* Infants under the age of 6 mo or adults over the age of 18

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 117175 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of collaborations between public and private entities to increase influenza vaccination in children 6 mos to 18 yrs in 10 intervention sites in 3 counties throughout the state of CO during the '10-11 & '11-12 flu seasons. | Up to 4 months post intervention (December 2012)
  Primary outcome measure is to increase the rate of receipt of ≥1 influenza vaccine during the post-intervention year(s) compared to the pre-intervention year among children 6 mos.-18 yrs in 10 intervention sites. Intervention practices will collaborate with their respective health departments and/or the VNA to help assist with the increase in volume of patients needing to be vaccinated against flu in the 2010-2011 and the 2011-2012 flu seasons. Billing data will be obtained from all 20 sites (intervention+control) and compared to evaluate the effectiveness of this collaboration.

SECONDARY OUTCOMES:
high-risk children receipt of influenza vaccination | baseline and intervention years 1 and 2
  increase in the rate of receipt of ≥1 influenza vaccine during the post-intervention year compared to the pre-intervention year among high-risk children
high-risk children fully immunized during influenza season | baseline and intervention years 1 and 2
  increase in the rate of high-risk children who were fully immunized during the season.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Children's Hospital
Locations (27):
- United States (27):
  - Tri County Health dept, Aurora, Colorado
  - Aurora Family Medicine, Aurora, Colorado
  - Forum Family Medicine, Aurora, Colorado
  - Premier Pediatrics, Brighton, Colorado
  - Indian Crest Pediatrics, Broomfield, Colorado
  - Centennial Pediatrics, Centennial, Colorado
  - Advanced Pediatrics, Centennial, Colorado
  - Greenwood Pediatrics, Centennial, Colorado
  - Pediatric Pathways, Centennial, Colorado
  - Pediatrics 5280, Centennial, Colorado
  - CIIS, Denver, Colorado
  - Hampden Medical Group, Englewood, Colorado
  - Family Practice Clinic, Fort Morgan, Colorado
  - Ft. Morgan Medical Group, Fort Morgan, Colorado
  - Haxtun Family Medicine, Haxtun, Colorado
  - Valley Medical Center, Julesburg, Colorado
  - Jefferson County Health dept, Lakewood, Colorado
  - Kids First, Lakewood, Colorado
  - Denver West Pediatrics, Lakewood, Colorado
  - Focus on Kids, Littleton, Colorado
  - Lone Tree Family Medicine, Lone Tree, Colorado
  - Crown Point Pediatrics, Parker, Colorado
  - Northeast County Health Dept, Sterling, Colorado
  - Mountain Land Pediatrics, Thornton, Colorado
  - Pediatrics West, Wheat Ridge, Colorado
  - Wray Clinic, Wray, Colorado
  - Yuma Clinic, Yuma, Colorado